CLINICAL TRIAL: NCT00880061
Title: An Open Label Dose Escalation Safety Study of Convection-Enhanced Delivery of IL13-PE38QQR in Patients With Progressive Pediatric Diffuse Infiltrating Brainstem Glioma and Supratentorial High-Grade Glioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090117; 09-N-0117
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2015-06-05

CONDITIONS: Brain Neoplasm; Glioma
Keywords: Diffuse Infiltrating Pontine Glioma; Supratentorial High Grade Glioma; Convection-Enhanced Delivery; Pediatric Brain Tumor; Brain Tumor; Glioma
MeSH Terms: conditions — Brain Neoplasms; Glioma | interventions — IL13-PE38

INTERVENTIONS:
Drug: IL13-PE38QQR

SUMMARY:
Background:

* Diffusely infiltrating pontine glioma (DIPG) or supratentorial high-grade glioma (HGG) are brain tumors that are often difficult to treat. It is very difficult to get chemotherapy agents to tumors in the brain, and researchers are looking for new methods to directly treat these types of cancer.
* IL-13 is an immune molecule normally occurring in the body. Patients with gliomas appear to have significant amounts of the IL-13 receptors in their brain tumors. An experimental drug, IL13-PE38QQR, combines a bacteria toxin with human IL-13 to allow the toxin to enter and destroy the tumor cell. Early clinical studies suggest this treatment may prolong survival of patients with these types of brain tumors.
* A technique called convection-enhanced delivery (CED) uses continuous pressure to push large molecules through the membranes protecting the brain to reach brain tumors. This technique can treat a tumor more directly than with traditional methods.

Objectives:

* To test the safety and feasibility of giving IL13-PE38QQR directly into regions of the brain in pediatric patients with DIPG or HGG, using CED.
* To determine the most appropriate dose of IL13-PE38QQR to treat DIPG or HGG.
* To determine the effects of this experimental therapy on the tumor.
* To evaluate the physical changes in the tumor before and after the therapy.

Eligibility:

* Patients who are less than 18 years of age and have been diagnosed with either DIPG or with supratentorial HGG that has not responded well to standard treatments.

Design:

* Patients will be admitted to the hospital and will receive a magnetic resonance imaging (MRI) scan to show the exact location of the tumor. A small plastic tube will be inserted surgically into the tumor area, and IL13-PE38QQR and a MRI contrast agent (gadolinium DTPA) will be infused into the area.
* MRI scans will monitor the process, and the tube will be removed after surgery.
* Doses will be adjusted over the course of the study.
* Patients who respond well to treatment may be eligible to receive a second infusion, no sooner than 4 weeks after the first treatment.
* Post-treatment visits:

Clinic visits 4 and 8 weeks after the treatment, and then every 8 weeks for up to 1 year.

* Physical examination with neurological testing, an MRI, and standard blood and urine tests.

DETAILED DESCRIPTION:
Objective: The primary purpose of this study is to test the safety and feasibility of giving a new experimental agent, called IL13-PE38QQR, directly into regions of the brain in patients with diffusely infiltrating pontine glioma (DIPG) or with recurrent or progressive supratentorial high-grade glioma (HGG) using a technique called convection-enhanced delivery or CED. CED uses continuous pressure to push large molecules through the membranes protecting the brain to reach brain tumors. At the same time, we can watch where the molecules go in the brain by attaching a tracer, gadolinium-DTPA, to the IL13-PE38QQR, which can then be seen in the brain with magnetic resonance imaging (MRI). Because we do not know the best dose to use in patients with DIPG or HGG, we will give increasing amounts of IL13-PE38QQR to small groups of patients with each type of brain tumor, known as a dose escalation study. Secondary purposes of this study include determining the effects of this experimental therapy on the tumor, and evaluating the physical changes in the tumor before and after the therapy.

Study Population: Twenty-right pediatric patients with recurrent or progressive DIPG or supratentorial HGG that have undergone standard treatment and who meet all the Inclusion and Exclusion Criteria may be enrolled. Eighteen patients will receive treatment; an additional ten patients may be screening failures or unevaluable.

Design: We propose a Phase I single institution, open label, dose escalation (doses of 0.125, 0.25 and 0.5 micrograms/ml), safety and tolerability study of IL13-PE38QQR infused via CED into patients with either DIPG (up to 9 patients) or recurrent HGG (up to 9 patients). IL13-PE38QQR will be administered to regions of tumor determined by radiographic findings. Escalating dose levels will be evaluated in the following dose cohorts (3 patients per Cohort): Cohort 1 = 0.125 micrograms/ml, Cohort 2 = 0.25 micrograms/ml and Cohort 3 = 0.5 micrograms/ml.

Outcome Measures: To assess the safety, tolerability and potential efficacy of CED of IL13-PE38QQR, we will use detailed clinical and radiographic examinations. These will be performed at baseline and on post-infusion days 1, 28 and 60. After post-infusion day 60, clinical and radiographic studies will then be performed every 8 weeks until imaging or clinical evidence of recurrence/progressive disease or new treatment is initiated.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age less than 18 years
* Diagnosis: recurrent or progressive:

  1. DIPG
  2. HGG
* Patients undergoing surgical resection must have measurable/evaluable disease prior to study entry.
* Histopathologic Diagnosis

  1. A histopathologic diagnosis is not required for patients with DIPG but a biopsy may be recommended if the patient has an atypical presentation or atypical findings on MR-imaging.
  2. Histopathologic confirmation for patients with HGG is required. If necrosis is suspected based on MR-imaging and Nuclear Medicine scans, biopsy or surgical resection for confirmation of disease progression may be required.
* Prior Therapy

  1. Patients must have received at least standard doses of radiation (i.e., greater than 54 Gy).
  2. Surgery/biopsy - Patients must be more than 2 weeks from any neurosurgical procedure and cleared by the Principal Investigator before undergoing CED.
  3. Radiation - Patients must be more than 4 weeks from last fraction of radiation to the target site
  4. Chemotherapy - Patients must not be on concurrent chemotherapy. The last dose of chemotherapy must be greater than 2 weeks prior to CED and the patient must have recovered from any toxic effects of prior therapy (to less than Grade 2 or baseline).
  5. Biologic therapy - Patients must be greater than 7 days from biologic therapy.
  6. Investigational therapy - Patients must be greater than 30 days from any investigational therapy.
* Patients must be healthy enough to tolerate surgery and general anesthesia in the opinion of the primary investigator. This includes, but is not limited to:

  1. Adequate baseline organ function, including an age-adjusted normal serum creatinine OR a creatinine clearance greater or equal to 60 mL/min/1.73m(2), total bilirubin less than 2 times the upper limit of normal (ULN) and direct bilirubin within normal limits. Patients with elevated SGPT (up to 5 times ULN) will be eligible if the elevation is attributed to steroid treatment.
  2. If neurological deficits are present, they must be stable for at least 1 week prior to registration.
* Patients must be able to undergo MR-imaging with gadolinium-based contrast administration (e.g. no ferrous-containing implants, no pacemakers, no allergy to contrast, etc).
* All patients or their legal guardians must sign a document of informed consent indicating their understanding of the investigational nature and the potential risks associated with this study. When appropriate, pediatric patients will be included in all discussions in order to obtain verbal and written assent.

EXCLUSION CRITERIA:

* Patients with an uncorrectable bleeding disorder
* Patients with multifocal or leptomeningeal disease
* Patients with signs of impending herniation or an acute intratumoral hemorrhage
* Patients on concurrent chemotherapy or biologic therapy for the treatment of their tumor
* Patients who are pregnant or breastfeeding, because of unknown effects of the study agent, the strong magnetic fields and Gadolinium containing contrast agents on the fetus; patients of child-bearing potential must be willing to practice an effective form of birth control, including abstinence, hormone therapy, intrauterine device, 2 barrier methods.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2009-04-07; Primary Completion 2015-06-05 (Actual); Study Completion 2015-06-05 (Actual)

PRIMARY OUTCOMES:
1) Feasibility of perfusing specific sites within the CNS with IL13-PE38QQR, administered concurrently with gd-DTPA, 2) Safety and tolerability of escalating doses of IL13-PE38QQR via CED to pediatric patient with DIPGs and HGGs

SECONDARY OUTCOMES:
Determine effect of IL13-PE38QQR on MRI tumor measurements, symptom improvement or worsening, changes on clinical exam, radiographic changes, steroid dosing, QOL testing and survival of pediatric patients with DIPG and recurrent HGG

CONTACTS AND LOCATIONS:
Overall Officials: John D Heiss, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Linabery AM, Ross JA. Trends in childhood cancer incidence in the U.S. (1992-2004). Cancer. 2008 Jan 15;112(2):416-32. doi: 10.1002/cncr.23169. PMID 18074355
- [Background] Packer RJ, Sutton LN, Goldwein JW, Perilongo G, Bunin G, Ryan J, Cohen BH, D'Angio G, Kramer ED, Zimmerman RA, et al. Improved survival with the use of adjuvant chemotherapy in the treatment of medulloblastoma. J Neurosurg. 1991 Mar;74(3):433-40. doi: 10.3171/jns.1991.74.3.0433. PMID 1847194
- [Background] Broniscer A, Gajjar A. Supratentorial high-grade astrocytoma and diffuse brainstem glioma: two challenges for the pediatric oncologist. Oncologist. 2004;9(2):197-206. doi: 10.1634/theoncologist.9-2-197. PMID 15047924
- [Derived] Robison NJ, Kieran MW. Diffuse intrinsic pontine glioma: a reassessment. J Neurooncol. 2014 Aug;119(1):7-15. doi: 10.1007/s11060-014-1448-8. Epub 2014 May 3. PMID 24792486
- [Derived] Chittiboina P, Heiss JD, Warren KE, Lonser RR. Magnetic resonance imaging properties of convective delivery in diffuse intrinsic pontine gliomas. J Neurosurg Pediatr. 2014 Mar;13(3):276-82. doi: 10.3171/2013.11.PEDS136. Epub 2014 Jan 10. PMID 24410126